CLINICAL TRIAL: NCT03178994
Title: The Study of Efficacy and Safety of 2% Ketoconazole Cream in Thai Females With Mild Degree of Post - Adolescence Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 317/60
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-07

CONDITIONS: Post - Adolescence Acne
Keywords: Post - adolescence acne; Topical 2% ketoconazole cream

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% ketoconazole cream (Experimental): 2% ketoconazole cream apply on face twice daily for 10 weeks.
  Interventions: Drug: 2% ketoconazole cream
- Placebo (Placebo Comparator): Hydrophilic cream (in-house preparation) apply on face twice daily for 10 weeks.
  Interventions: Drug: Hydrophilic Cream

INTERVENTIONS:
Drug: 2% ketoconazole cream — 2% ketoconazole cream applies twice daily
  Arms: 2% ketoconazole cream
Drug: Hydrophilic Cream — Hydrophilic cream (in-house preparation) applies twice daily
  Arms: Placebo

SUMMARY:
To study efficacy (total numbers of acne reduction) and safety of 2% Ketoconazole cream in Thai females with Mild degree Post-Adolescence acne comparing with placebo for a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycle with mild degree of post - adolescence acne
* agree to stop topical and systemic medication for acne treatment for 2 and 4 weeks respectively.

Exclusion Criteria:

* Pregnancy or lactation
* Other active rashes on faces.
* Allergic to ketoconazole or other ingredients of preparation.
* Signs of hyperandrogenism
* Taking anti-androgenic medications.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Total numbers of acne reduction | 10 weeks
  the difference of acne count (total numbers of acne before treatment - total numbers of acne after treatment)

SECONDARY OUTCOMES:
Proportion of patients who achieve clear or almost clear after treatment | 10 weeks
  clear or almost clear scored by Adult Female Acne Scoring Tool

CONTACTS AND LOCATIONS:
Overall Officials: Chanat Kumtornrut, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Medicine, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided